CLINICAL TRIAL: NCT01695291
Title: A Randomized, Placebo-controlled Trial of Minocycline Added to Serotonin Reuptake Inhibitors in Pediatric OCD: Examining the Effects on Clinical Symptoms and on Brain Glutamate Levels Using MRS Imaging
Brief Title: Novel Medication Strategies Targeting Brain Mechanisms in Pediatric OCD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Helen Blair Simpson, Research Chief, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6574; R34MH095502-03 (NIH)
Record Dates: First submitted 2012-09-21; First posted 2012-09-27 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive compulsive disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants randomized to placebo will receive pills that are identical in appearance to the study drug but contain no active medication.
  Interventions: Other: Placebo
- Minocycline Augmentation (Experimental): Those randomized to minocycline will receive approximately 2 mg/kg/day, the FDA-approved dose for minocycline (minimum 50 mg/day and maximum 200 mg/day). After randomization, participants will receive child proofed bottles that contain enough study medication until the next visit with an additional 3 days coverage in case of scheduling issues. All participants will have a minocycline level drawn at week 12 to confirm treatment adherence. Minocycline is FDA-approved in those ages 8 and above for treatment of infections and acne and has a favorable risk-benefit profile.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Participants randomized to minocycline will receive approximately 2 mg/kg/day, the FDA-approved dose for minocycline. Participants will take either minocycline or pill placebo for 12 weeks.
  Other Names: Minomycin, Minocin, Arestin, Aknemin, Solodyn and Dynacin
  Arms: Minocycline Augmentation
Other: Placebo — A placebo pill will be administered twice a day (BID) for 12 weeks.
  Arms: Placebo

SUMMARY:
This study will examine the feasibility and potential efficacy of augmenting SRIs with minocycline. The study will assess whether the addition of minocycline leads to measurable changes in striatal glutamate (Glu) levels. This study will recruit up to 45 youth ages 8-20 diagnosed with clinically significant OCD who have demonstrated no more than minimal response to SRI treatment and are currently on a stable dose of SRI medication for at least 12 weeks. Participants will be randomized to receive either 12 weeks of minocycline treatment or pill placebo. Randomization will be 2:1 so that 2 of 3 participants receive minocycline. Screening for eligibility will take place for 1-4 weeks. Participants will undergo magnetic resonance spectroscopy (MRS) scans to measure striatal Glu levels prior to randomization, and again immediately following the treatment period. During the treatment period, participants will meet initially weekly and then every other week with the study psychiatrist. All participants will be offered three months of open medication treatment following participation. The clinical trial will only be conducted at the New York State Psychiatric Institute (NYSPI) and the MRS scans may be conducted at Weill Cornell Medical Center or NYSPI.

DETAILED DESCRIPTION:
Please see the brief summary for study description.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ages of 8-20 at the time of consent
* Participants must weigh at least 25kg
* Participants and a parent/guardian must be able to read and understand English
* Participants must meet diagnostic criteria for obsessive-compulsive disorder with score ≥ 16 on the Children's Yale-Brown Obsessive Compulsive Scale (CYBOCS)
* Participants must be on stable dose of serotonin reuptake inhibitor (SRI) medication, and must have had a minimal adequate trial of SRI medication
* Report of at least minimal, but not full, response to current SRI medication to warrant ongoing SRI treatment
* For participants younger than 18, written informed assent by the participant and consent by the parent. For participants 18 and older, written consent by the participant and permission for legal guardian/parent to provide information

Exclusion Criteria:

* Lifetime diagnosis of: psychotic disorder, bipolar disorder, eating disorder, pervasive developmental disorder, mental retardation, or substance/alcohol dependence
* Current diagnosis of major depressive disorder, Tourette's/Tic Disorder, or substance/alcohol abuse
* Positive urine screen for illicit drugs
* Medical or psychiatric conditions that would make participation in the study unsafe
* Active suicidal ideation
* Females who are using hormonal birth control
* Presence of metallic device or dental braces incompatible with MRS
* Intelligence quotient (IQ) <80
* OCD patients with primary symptoms of hoarding (determined by CYBOCS checklist)
* Current or past diagnosis of pediatric autoimmune neuropsychiatric disorders associated with streptococcus (PANDAS)
* Individuals who are currently receiving Exposure and Response Prevention therapy and are in the acute phase of treatment.
* Documented history of hypersensitivity or intolerance to tetracycline antibiotics
* Use of medications that are contra-indicated with minocycline (e.g., concomitant use of antacids, iron, calcium, magnesium, aluminum, zinc salts as they impair minocycline absorption; of anti-coagulant drugs as minocycline has been shown to depress plasma prothrombin activity; of other antibiotics or Accutane due to the rare side effect of pseudotumor cerebri)
* Inability of participant or parent/guardian to read or understand English

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moira A Rynn, M.D., Principal Investigator — Columbia University/NYSPI
Locations (2):
- United States (2):
  - Weill Cornell Medical Center, New York, New York
  - New York State Psychiatric Institute, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Minocycline Augmentation
Started | 10 | 21
Completed | 8 | 14
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants randomized to placebo will receive pills that are identical in appearance to the study drug but contain no active medication.
  Placebo: A placebo pill will be administered BID for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Minocycline Augmentation | Total
Number analyzed (Participants) | 10 | 21 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 16 | 24
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 20 | 28
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 19 | 24
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 21 | 31

OUTCOME MEASURES:

1. Primary Outcome: Yale-Brown Obsessive Compulsive Scale, Child Version (CYBOCS)
Description: The Yale-Brown Obsessive Compulsive Scale, Child Version (CYBOCS) is a semi-structured measure of Obsessive-Compulsive Disorder (OCD) severity with excellent inter-rater reliability, internal consistency, and test-retest reliability. It is validated in those starting at age 7 and used in studies up to age 20. The CYBOCS differs from the adult YBOCS only in its use of simpler language. The total CYBOCS score ranges from 0 to 40, with higher scores indicating more severe symptomatology.
Time Frame: Change from Baseline at 4, 8, and 12 weeks
Population: Due to the early-termination of some participants, not all completed the CYBOCS at Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Minocycline Augmentation
Number analyzed (Participants) | 10 | 21
units on a scale
  Baseline | 28.20 (3.79) | 29.0 (3.49)
  Week 4: number analyzed (Participants) | 9 | 18
  Week 4 | 26.67 (4.69) | 27.11 (5.61)
  Week 8: number analyzed (Participants) | 9 | 17
  Week 8 | 25.33 (5.22) | 25.47 (5.77)
  Week 12: number analyzed (Participants) | 9 | 17
  Week 12 | 26.44 (5.10) | 25.59 (6.39)

2. Secondary Outcome: Striatal Glutamate Level Measured by Magnetic Resonance Spectroscopy (MRS).
Description: The change in striatal glutamate level will be assessed.
Time Frame: Change from Baseline at 12 weeks
Population: Due to the early-termination of some participants, not all completed MRS at Week 12
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Placebo | Minocycline Augmentation
Number analyzed (Participants) | 9 | 17
Arbitrary Units
  Baseline | 44.49 (6.76) | 43.96 (9.18)
  Week 12: number analyzed (Participants) | 8 | 14
  Week 12 | 42.97 (8.25) | 39.35 (6.47)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Minocycline Augmentation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/10 | 5/21
Other Adverse Events (participants affected / at risk) | 10/10 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Minocycline Augmentation (N=21)
Hospitalization (Psychiatric disorders) | 0 | 2 — For increased hostility and threatening behaviors (N=1) and for worsening OCD symptoms (N=1)
Drug Rash (Skin and subcutaneous tissue disorders) | 0 | 1 — Drug rash requiring prednisone treatment
Significant esophagitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Worsening of OCD symptoms and an interrupted suicide attempt (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Minocycline Augmentation (N=21)
Irritable or bad mood (Psychiatric disorders) | 2 | 5
Angry or hostile (Psychiatric disorders) | 1 | 6
Sad or low mood (Psychiatric disorders) | 4 | 7
Lack of interest (Psychiatric disorders) | 4 | 6
Feeling shutdown (Psychiatric disorders) | 4 | 3
Mood swings (Psychiatric disorders) | 3 | 5
Anxious, tense, uptight (Psychiatric disorders) | 2 | 6
Lack of self-control/impulsive (Psychiatric disorders) | 4 | 1
Trouble paying attention (Psychiatric disorders) | 3 | 3
Racing thoughts (Psychiatric disorders) | 4 | 3
Can't sit or stand still (Psychiatric disorders) | 4 | 7
Tired/fatigued (Psychiatric disorders) | 5 | 5
Sleep too much (Psychiatric disorders) | 2 | 8
Trouble falling or staying asleep (Psychiatric disorders) | 3 | 4
Lost weight (Metabolism and nutrition disorders) | 1 | 1
Dry mouth (General disorders) | 1 | 1
More thirsty (General disorders) | 1 | 2
Feeling hungry (Metabolism and nutrition disorders) | 1 | 2
Gained weight (Metabolism and nutrition disorders) | 1 | 0
Muscles weak (Musculoskeletal and connective tissue disorders) | 1 | 2
Pimples or acne (Skin and subcutaneous tissue disorders) | 1 | 0
Heart racing or skipping beats (Cardiac disorders) | 0 | 3
Stomach ache or cramps (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Headache (General disorders) | 1 | 4
Less hungry (Metabolism and nutrition disorders) | 0 | 2
Dizzy or light-headed (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT01695291/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT01695291/SAP_001.pdf